CLINICAL TRIAL: NCT01947868
Title: A Prospective, Non-interventional Evaluation of Symptoms Improvement of First-Line Therapy of EGFR Tyrosine Kinase Inhibitor in Advanced NSCLC Patients With Positive EGFR Mutation - the SMILE Study
Brief Title: Evaluation of Symptoms Improvement in NSCLC Patients With First-Line Therapy of EGFR Tyrosine Kinase Inhibitor
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OTW-ATC-2013/1
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — no biospecimen collected
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an open-label, non-interventional, single-arm, multicenter study in a real-world population to assess the clinically symptom improvement and quality of life (QoL) in patients with locally advanced or metastatic NSCLC and positive EGFR mutation who receive EGFR-TKIs as the first-line treatment.

The Primary Objective is to estimate symptom improvement rates in patients with locally advanced or metastatic NSCLC and positive EGFR mutation who receive EGFR-TKIs as the first-line treatment. A clinically meaningful improvement is defined as an increase from baseline of 2 or more points for LCS (Lung Cancer Scales) at Week 4.

DETAILED DESCRIPTION:
The Secondary Objectives are:

1. To estimate symptom improvement rates at weeks 2 and 12
2. To estimate mean change from baseline in overall QoL scores using the FACT-L instrument and LCS score at Week 2, 4 and 12.
3. To estimate the proportion of patients exhibiting an LCS change of 7 points or more at weeks 2, 4 and 12.
4. Subgroup information of symptom improvement rate, QoL and disease-related symptom scores by gender, smoking status, smoking pattern, WHO performance, number of metastatic sites, female/never smokers and patients with COPD at week 2, week 4 and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with symptomatic, locally advanced or metastatic (stage IIIb/IV) NSCLC.
* Patients who are positive for EGFR mutation
* Patients with a prescription of EGFR-TKI as their first-line treatment

Exclusion Criteria:

- Involvement in any planning and/or conduct of the clinical trial.

Ages: 20 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced NSCLC patients who will be treated as first line treatment with EGFR-TKI
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients demonstrating a clinically meaningful improvement post 4 weeks of EGFR-TKI therapy defined as an increase in LCS ≥ 2 points from baseline. | 15 months
  LCS is Lung Cancer Scale

SECONDARY OUTCOMES:
The proportion of patients demonstrating a clinically meaningful improvement post 2 weeks and 12 weeks of EGFR-TKI therapy as defined as an increase in LCS ≥ 2 points from baseline. | 15 months
Mean change from baseline to Week 2, 4 and 12 in FACT-L, TOI and LCS. | 15 months
  FACT-L is Functional Assessment of Cancer Therapy-Lung questionnaire. TOI is Treatment Outcome Index. LCS is Lung Cancer Scale.
The proportion of patients demonstrating a clinically meaningful improvement post 2, 4 and 12 weeks of EGFR-TKI therapy as defined as an increase in LCS ≥ 7 points from baseline. | 15 months
  LCS is Lung Cancer Scale
Descriptive statistics in improvement rate (defined as LCS ≥ 2 points changed from baseline), QoL and disease-related symptom scores at week 2,4 and 12 and summarized by gender, smoking status, smoking pattern, WHO performance status, etc | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Te-Chun Hsia, Principal Investigator — 886422062121
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- See also: NIS-OTW-ATC-2013_1_CSR_Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1894&filename=NIS-OTW-ATC-2013_1_CSR_Synopsis.pdf